CLINICAL TRIAL: NCT00669214
Title: A Phase IV Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of 1.0 mg/kg Efalizumab in Adult Patients With Moderate to Severe Plaque Psoriasis With Involvement of the Scalp
Brief Title: A Study to Evaluate the Safety and Efficacy of Efalizumab in Adult Patients With Moderate to Severe Plaque Psoriasis With Involvement of the Scalp
Acronym: SCALP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACD4412n
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis
Keywords: Raptiva; Moderate plaque psoriasis; Severe plaque psoriasis; Scalp
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Efalizumab (Experimental)
  Interventions: Drug: efalizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: efalizumab — All patients received a conditioning dose of efalizumab 0.7 mg/kg subcutaneously (SC) on Day 0, followed by 11 weekly doses of 1.0 mg/kg SC beginning on Day 7. After 12 weeks of blinded treatment, all patients continued into the open-label treatment period from Day 84 (Week 12) through Day 168 (Week 24).
  Other Names: Raptiva
  Arms: Efalizumab
Drug: placebo — All patients received a conditioning dose of placebo equivalent SC on Day 0, followed by 11 weekly doses of placebo SC beginning on Day 7. After 12 weeks of blinded treatment, all patients continued into the open-label efalizumab treatment period from Day 84 (Week 12) through Day 168 (Week 24).
  Arms: Placebo

SUMMARY:
This was a Phase IV randomized, double-blind, placebo-controlled study designed to evaluate the safety and efficacy of subcutaneous efalizumab in adult patients (18 years of age and older) with chronic moderate to severe plaque psoriasis with involvement of the scalp who had no previous exposure to efalizumab. The study consisted of a screening period, a double-blind treatment period, an open-label treatment period, and an observation/follow-up period. The study enrolled 100 patients. 11 patients were excluded from all analyses because of data issues.

DETAILED DESCRIPTION:
* Baselines for Raptiva group and placebo group at Day 84 are the same. The baseline is Day 0.
* Baselines for Raptiva group and placebo group at Day 168 are different. The baseline for Raptiva group at Day 168 is Day 0, but the baseline for Placebo group at Day 168 is Day 84

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) documents
* Be aged 18 years or older
* Have chronic (6 months or greater) moderate to severe plaque psoriasis with involvement of the scalp
* Have a whole body Physician's Global Assessment (PGA) rating of moderate (3) or severe (4) for psoriasis
* Have a scalp surface area affected by plaque psoriasis of 30% or more, assessed using Psoriasis Scalp Severity Index (PSSI)
* Have at least one of three clinical signs involving the scalp (erythema, induration, and desquamation) be rated as at least moderate (2) with the other two rated as at least slight (1) using PSSI
* Be a candidate for systemic therapy in the opinion of the investigator
* Be naive to efalizumab treatment
* For women of childbearing potential, must be willing to use a method of contraception acceptable to the investigator to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study and for 6 weeks after the last dose of efalizumab

Exclusion Criteria:

* Have had previous exposure to efalizumab or a history of hypersensitivity to any of its components
* Are using any excluded therapy
* Have a history of drug or alcohol abuse in the past five years
* Have a history in the past 5 years of a serious infection or currently have an ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* Have any history of opportunistic infections (e.g., systemic fungal infections, parasites)
* Are seropositive for hepatitis B antigen, hepatitis C antibody, or human immunodeficiency virus (HIV)
* Have a history of active tuberculosis or are currently undergoing treatment for tuberculosis, including latent tuberculosis with isoniazid
* Have the presence or history of malignancy within the past 5 years, including lymphoproliferative disorders
* Are pregnant or breastfeeding
* Have a diagnosis of hepatic cirrhosis, regardless of cause or severity
* Have a history in the last 5 years of thrombocytopenia
* Have a history in the last 5 years of hemolytic anemia or any other clinically significant anemia
* Have been exposed to any experimental and/or unapproved drugs or treatments within 30 days or 5 half-lives, whichever is longer, before the screening visit
* Have been vaccinated with a live virus or live bacteria within the 14 days before the first dose of efalizumab
* Have any medical condition that, in the judgment of the investigator, would jeopardize the patient's safety following exposure to study drug (efalizumab or placebo equivalent) or would significantly interfere with the patient's ability to comply with the provisions of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Caro, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: All patients received a conditioning dose of placebo equivalent subcutaneously (SC) on Day 0, followed by 11 weekly doses of placebo SC beginning on Day 7. After 12 weeks of blinded treatment, all patients continued into the open-label efalizumab treatment period from Day 84 (Week 12) through Day 168 (Week 24).
Period: Double-Blind Treatment Period (Week 12)
Arm/Group | Placebo | Efalizumab
Started | 27 | 62
Completed | 22 | 55
Not Completed | 5 | 7
Period: Open-Label Treatment Period (Week 24)
Arm/Group | Placebo | Efalizumab
Started | 22 | 55
Completed | 18 | 46
Not Completed | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Efalizumab | Total
Number analyzed (Participants) | 27 | 62 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.78 (16.53) | 43.16 (13.46) | 43.04 (14.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 30 | 39
  Male | 18 | 32 | 50

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieved a ≥ 75% Decrease in Psoriasis Scalp Severity Index (PSSI) Score at 12 Weeks
Description: Proportion of patients who achieved a ≥ 75% decrease in PSSI score at 12 weeks (Day 84) relative to baseline. The PSSI assessed: 1) extent of scalp psoriasis (i.e., percentage of area involved), which was scored from 1 to 6, where 1 = <10% and 6 = 90-100%); and 2) clinical signs (erythema, induration, and desquamation), which were scored from 0 to 4, where 0 = Absent and 4 = Severest possible). The sum of the separate scores for erythema, induration, and desquamation was multiplied by the score for the involved area. The PSSI score range was therefore 0-72.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population. If PSSI at Day 84 was missing for a patient who discontinued before the final scheduled dose, the patient was considered a treatment failure (nonresponder) for analysis. If PSSI at Day 84 was missing for a patient who completed treatment, the last available PSSI from the treatment period was used for analysis.
Measure: Number; unit: Proportion of patients
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 27 | 62
Proportion of patients | 0.111 | 0.274
Statistical Analysis 1: Comparison: Placebo vs Efalizumab; Test type: Superiority or Other; p = 0.1054, Fisher Exact; The p-value was based on the Fisher exact test for a 2x2 contingency table; Difference in proportion = 0.163, 95% CI [-0.063 to 0.393]

2. Secondary Outcome: Proportion of Patients Who Achieved a ≥ 75% Decrease in PSSI Score at 24 Weeks
Description: Proportion of patients who achieved a ≥ 75% decrease in PSSI score at 24 weeks (Day 168) relative to baseline. The PSSI assessed: 1) extent of scalp psoriasis (i.e., percentage of area involved), which was scored from 1 to 6, where 1 = <10% and 6 = 90-100%); and 2) clinical signs (erythema, induration, and desquamation), which were scored from 0 to 4, where 0 = Absent and 4 = Severest possible). The sum of the separate scores for erythema, induration, and desquamation was multiplied by the score for the involved area. The PSSI score range was therefore 0-72.
Time Frame: Week 24
Population: ITT population. If PSSI at Day 168 was missing for a patient who discontinued before the final scheduled open-label dose, the patient was considered a treatment failure (nonresponder) for analysis. If PSSI at Day 168 was missing for a patient who completed the Day 161 dose, the last available PSSI was used for analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 22 | 62
Proportion of patients | 0.273 [0.107 to 0.502] | 0.323 [0.209 to 0.453]

3. Secondary Outcome: Proportion of Patients Who Achieved a ≥ 50% Decrease in PSSI Score at 12 Weeks
Description: Proportion of patients who achieved a ≥ 50% decrease in PSSI score at 12 weeks (Day 84) relative to baseline. The PSSI assessed: 1) extent of scalp psoriasis (i.e., percentage of area involved), which was scored from 1 to 6, where 1 = <10% and 6 = 90-100%); and 2) clinical signs (erythema, induration, and desquamation), which were scored from 0 to 4, where 0 = Absent and 4 = Severest possible). The sum of the separate scores for erythema, induration, and desquamation was multiplied by the score for the involved area. The PSSI score range was therefore 0-72.
Time Frame: Week 12
Population: ITT population. If PSSI at Day 84 was missing for a patient who discontinued before the final scheduled dose, the patient was considered a treatment failure (nonresponder) for analysis. If PSSI at Day 84 was missing for a patient who completed treatment, the last available PSSI from the treatment period was used for analysis.
Measure: Number; unit: Proportion of patients
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 27 | 62
Proportion of patients | 0.296 | 0.452
Statistical Analysis 1: Comparison: Placebo vs Efalizumab; Test type: Superiority or Other; p = 0.2404, Fisher Exact; The p-value was based on the Fisher exact test for a 2x2 contingency table; Difference in proportion = 0.155, 95% CI [-0.072 to 0.388]

4. Secondary Outcome: Proportion of Patients Who Achieved a ≥ 50% Decrease in PSSI Score at 24 Weeks
Description: Proportion of patients who achieved a ≥ 50% decrease in PSSI score at 24 weeks (Day 168) relative to baseline. The PSSI assessed: 1) extent of scalp psoriasis (i.e., percentage of area involved), which was scored from 1 to 6, where 1 = <10% and 6 = 90-100%); and 2) clinical signs (erythema, induration, and desquamation), which were scored from 0 to 4, where 0 = Absent and 4 = Severest possible). The sum of the separate scores for erythema, induration, and desquamation was multiplied by the score for the involved area. The PSSI score range was therefore 0-72.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 22 | 62
Proportion of patients | 0.455 [0.244 to 0.678] | 0.500 [0.370 to 0.630]

5. Secondary Outcome: Proportion of Patients Who Achieved a Whole Body (Including Scalp) Physician's Global Assessment (PGA) Rating of Clear (0), Almost Clear (1), or Mild (2) at 12 Weeks
Description: Proportion of patients who achieved a whole body (including scalp) PGA rating of 0, 1, or 2 at 12 weeks (Day 84)
  Physician's Global Assessment (PGA) scale:
  0: Clear. No signs of plaque psoriasis.
  1. Almost clear. Just perceptible erythema and just perceptible scaling.
  2. Mild disease. Light pink erythema with minimal scaling.
  3. Moderate disease. Dull red, clearly distinguishable erythema with diffuse scaling, some thickening.
  4. Severe disease. Deep/dark red erythema with clearly obvious and diffuse scaling and thickening.
Time Frame: Week 12
Population: ITT population. If PGA rating at Day 84 was missing for a patient who discontinued before the final scheduled dose, the patient was considered a treatment failure (nonresponder) for analysis. If PGA rating at Day 84 was missing for a patient who completed treatment, the last available PGA rating from the treatment period was used for analysis.
Measure: Number; unit: Proportion of patients
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 27 | 62
Proportion of patients | 0.111 | 0.339
Statistical Analysis 1: Comparison: Placebo vs Efalizumab; Test type: Superiority or Other; p = 0.0366, Fisher Exact; The p-value was based on the Fisher exact test for a 2x2 contingency table; Difference in proportion = 0.228, 95% CI [0.003 to 0.452]

6. Secondary Outcome: Proportion of Patients Who Achieved a Whole Body (Including Scalp) PGA Rating of Clear (0), Almost Clear (1), or Mild (2) at 24 Weeks
Description: Proportion of patients who achieved a whole body (including scalp) PGA rating of 0, 1, or 2 at 24 weeks (Day 168) For details on the PGA scale, refer to the Secondary Outcome Measure Description for 12 weeks.
Time Frame: Week 24
Population: ITT population. If PGA rating at Day 168 was missing for a patient who discontinued before the final scheduled open-label dose, the patient was considered a treatment failure (nonresponder) for analysis. If PGA rating at Day 168 was missing for a patient who completed the Day 161 dose, the last available PGA rating was used for analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 22 | 62
Proportion of patients | 0.545 [0.322 to 0.756] | 0.387 [0.266 to 0.519]

7. Secondary Outcome: Mean Change in Scalpdex Score at 12 Weeks
Description: Mean change in Scalpdex score at 12 weeks (Day 84) relative to baseline. The Scalpdex point scoring scale ranges from 1=NEVER, 2='RARELY', 3='SOMETIMES', 4='OFTEN' and 5='ALL THE TIME'.
Time Frame: The two time points for Mean Change in Scalpdex Score at 12 Weeks are Day 0 and Day 84
Population: ITT population. If Scalpdex at Day 84 was missing for a patient who discontinued before the final scheduled dose, the patient was not included in the analysis. If Scalpdex at Day 84 was missing for a patient who completed treatment, the last available Scalpdex from the treatment period was used for analysis.
Measure: Mean (Standard Deviation); unit: Points on Scalpdex
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 22 | 55
Points on Scalpdex
  Baseline Score | 63.91 (15.40) | 67.83 (13.88)
  Week 12 Change from Baseline | 6.82 (7.76) | 10.15 (13.56)
Statistical Analysis 1: Comparison: Placebo vs Efalizumab; Test type: Superiority or Other; p = 0.1816, Student T-test; Difference in mean change from Day 0 = 3.33, 95% CI [-2.811 to 9.471]

8. Secondary Outcome: Mean Change in Scalpdex Score at 24 Weeks
Description: Mean change in Scalpdex score at 24 weeks (Day 168) relative to baseline. The Scalpdex point scoring scale ranges from 1=NEVER, 2='RARELY', 3='SOMETIMES', 4='OFTEN' and 5='ALL THE TIME'.
Time Frame: Week 24
Population: ITT population. If Scalpdex at Day 168 was missing for a patient who discontinued before the final scheduled dose, the patient was not included in the analysis. If Scalpdex at Day 168 was missing for a patient who completed the Day 161 dose, the last available Scalpdex was used for analysis.
Measure: Mean (Standard Deviation); unit: Points on Scalpdex
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 18 | 47
Points on Scalpdex
  Baseline Score | 63.91 (15.40) | 67.83 (13.88)
  Week 24 Change from Baseline | 7.81 (9.80) | 13.26 (14.02)

9. Secondary Outcome: Mean Change in a Visual Analog Scale (VAS) of Scalp Itch at 12 Weeks
Description: Mean change in VAS of patient-reported scalp itch at 12 weeks (Day 84) relative to baseline. The Visual Analog Scale (VAS) of patient-reported scalp itch measured the severity of a patient's scalp itch on a scale of 0 to 10, where 0 was "no itching," 5 was "moderate itching," and 10 was "severe itching."
Time Frame: Week 12
Population: ITT population. If VAS at Day 84 was missing for a patient who discontinued before the final scheduled dose, the patient was not included in the analysis. If VAS at Day 84 was missing for a patient who completed treatment, the last available VAS from the treatment period was used for analysis.
Measure: Mean (Standard Deviation); unit: Points on VAS
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 22 | 54
Points on VAS
  Baseline Scale | 6.81 (2.34) | 7.47 (2.24)
  Week 12 Change from Baseline | 1.00 (1.95) | 2.19 (2.91)
Statistical Analysis 1: Comparison: Placebo vs Efalizumab; Test type: Superiority or Other; p = 0.0435, Student T-test; Difference in mean change from Day 0 = 1.19, 95% CI [-0.161 to 2.532]

10. Secondary Outcome: Mean Change in VAS of Patient-reported Scalp Itch at 24 Weeks
Description: Mean change in VAS of patient-reported scalp itch at 24 weeks (Day 168) relative to baseline. The Visual Analog Scale (VAS) of patient-reported scalp itch measured the severity of a patient's scalp itch on a scale of 0 to 10, where 0 was "no itching," 5 was "moderate itching," and 10 was "severe itching."
Time Frame: Week 24
Population: ITT population. If VAS at Day 168 was missing for a patient who discontinued before the final scheduled dose, the patient was not included in the analysis. If VAS at Day 168 was missing for a patient who completed the Day 161 dose, the last available VAS was used for analysis.
Measure: Mean (Standard Deviation); unit: Points on VAS
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 18 | 46
Points on VAS
  Baseline Points | 6.81 (2.34) | 7.47 (2.24)
  Week 24 Change from Baseline | 2.06 (3.61) | 3.07 (3.09)

11. Secondary Outcome: Mean Change in Percentage of Whole Body (Including Scalp) Body Surface Area (BSA) Affected by Psoriasis at 12 Weeks
Description: Mean change in percentage of whole body (including scalp) BSA affected by psoriasis at 12 weeks (Day 84) relative to baseline. BSA was assessed by percentage of sites affected per body segment (head, trunk, and limbs). Investigators were instructed to use the "rule of palm" to estimate lesional skin BSA (1% BSA = palm to first interphalangeal joint).
Time Frame: Week 12
Population: ITT population. N's reflect patients who received at least one dose of study drug or placebo in the double-blind treatment period.
Measure: Mean (Standard Deviation); unit: Pecentage of BSA
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 22 | 56
Pecentage of BSA
  Baseline BSA | 14.74 (15.48) | 19.61 (18.51)
  Week 12 Change from Baseline | 2.00 (5.65) | 6.43 (10.30)
Statistical Analysis 1: Comparison: Placebo vs Efalizumab; Test type: Superiority or Other; p = 0.0224, Wilcoxon rank sum

12. Secondary Outcome: Mean Change in Percentage of Whole Body (Including Scalp) BSA Affected by Psoriasis at 24 Weeks
Description: Mean change in percentage of whole body (including scalp) BSA affected by psoriasis at 24 weeks (Day 168) relative to baseline. BSA was assessed by percentage of sites affected per body segment (head, trunk, and limbs). Investigators were instructed to use the "rule of palm" to estimate lesional skin BSA (1% BSA = palm to first interphalangeal joint).
Time Frame: Week 24
Population: ITT population. N's reflect patients who received at least one dose of study drug in the open-label period.
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Placebo | Efalizumab
Number analyzed (Participants) | 18 | 48
Percentage of BSA
  Baseline BSA | 14.74 (15.48) | 19.61 (18.51)
  Week 24 Change from Baseline | 4.53 (6.53) | 7.53 (12.59)

ADVERSE EVENTS:
Time Frame: Double-blind (12 weeks), open-label (24 weeks), and follow-up. Patients entered each period as follows: Double-blind: placebo n = 27; efalizumab n = 62 Open-label: placebo n = 22; efalizumab n = 55 Follow-up: placebo n = 18; efalizumab n = 48
Groups:
- Placebo: Double-Blind Period: All patients received a conditioning dose of placebo equivalent SC on Day 0, followed by 11 weekly doses of placebo SC beginning on Day 7. After 12 weeks of blinded treatment, all patients continued into the open-label efalizumab treatment period from Day 84 (Week 12) through Day 168 (Week 24).
- Efalizumab: Double-Blind Period: All patients received a conditioning dose of efalizumab 0.7 mg/kg subcutaneously (SC) on Day 0, followed by 11 weekly doses of 1.0 mg/kg SC beginning on Day 7. After 12 weeks of blinded treatment, all patients continued into the open-label treatment period from Day 84 (Week 12) through Day 168 (Week 24).
Arm/Group | Placebo: Double-Blind Period | Efalizumab: Double-Blind Period | Placebo: Open-Label Period | Efalizumab: Open-Label Period | Placebo: Follow-Up Period | Efalizumab: Follow-Up Period
Serious Adverse Events (participants affected / at risk) | 1/27 | 1/62 | 0/22 | 1/55 | 0/18 | 2/48
Other Adverse Events (participants affected / at risk) | 11/27 | 32/55 | 11/22 | 22/55 | 3/18 | 15/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Double-Blind Period (N=27) | Efalizumab: Double-Blind Period (N=62) | Placebo: Open-Label Period (N=22) | Efalizumab: Open-Label Period (N=55) | Placebo: Follow-Up Period (N=18) | Efalizumab: Follow-Up Period (N=48)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Double-Blind Period (N=27) | Efalizumab: Double-Blind Period (N=55) | Placebo: Open-Label Period (N=22) | Efalizumab: Open-Label Period (N=55) | Placebo: Follow-Up Period (N=18) | Efalizumab: Follow-Up Period (N=48)
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Injection site hematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cyst rupture (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cat scratch disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Full blood count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Colonoscopy (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 10 | 3 | 1 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 5 | 2 | 3 | 0 | 2
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0
Nephrolithiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Since the completion of this study, efalizumab has been voluntarily withdrawn from the U.S. market because of a safety issue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.